CLINICAL TRIAL: NCT03142022
Title: Sleep-disordered Breathing After Solid Organ Transplantation
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S53746
Record Dates: First submitted 2016-09-27; First posted 2017-05-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Lung Transplantation; Sleep-disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SDB and lung transplantation: Polysomnography at 1 year after lung transplantation.
  Interventions: Other: No intervention - Diagnostic polysomnography at 1 year after lung transplantation

INTERVENTIONS:
Other: No intervention - Diagnostic polysomnography at 1 year after lung transplantation

SUMMARY:
Sleep-disordered breathing (SDB) describes a group of disorders in which partial or complete cessation of breathing occurs many times throughout the night, resulting in daytime sleepiness or fatigue that interferes with a person's ability to function and reduces quality of life. Transplantation has become an important treatment modality for end-stage organ failure. Transplant recipients are now living longer and, hence, develop chronic adverse medical conditions. Furthermore, transplantation is associated with weight gain. Despite the high prevalence of poor sleep and cardiovascular conditions among transplant patients, SDB is not well studied in these patients.

DETAILED DESCRIPTION:
The primary research objective is to evaluate the prevalence, incidence and type (central or obstructive) of SDB in patients after lung transplantation.

Secondary research objectives are the evaluation of correlations between severity of SDB and clinical findings (weight, medical therapy, heart function, lung function, renal function, graft failure, …). Furthermore, the investigators will evaluate the relationship between SDB and cardiovascular morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients 1 year after lung transplantation

Exclusion Criteria:

* Refusal of PSG
* Medical contra-indication to perform PSG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 1 year after lung transplantation are systematically evaluated by polysomnography.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with SDB and type (central or obstructive) of SDB | 1 year after lung transplantation
  Prevalence of different types of SDB after lung transplantation

SECONDARY OUTCOMES:
Echocardiography | 1 year after lung transplantation
  Correlations between SDB and heart function
Lung function measurement | 1 year after lung transplantation
  Correlations between SDB and lung function
Blood analysis | 1 year after lung transplantation
  Correlations between SDB and renal function
24h blood pressure | 1 year after lung transplantation
  Evaluation of relationship between hypertension and SDB

CONTACTS AND LOCATIONS:
Overall Officials: Dries Testelmans, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No